CLINICAL TRIAL: NCT06239298
Title: A Multi-center, Open, Dose Exploration and Dose Expansion Phase I/II Study of ZG005 Combined With Donafenib Tosilate Tablets in Patients With Advanced Solid Tumor
Brief Title: A Study of ZG005 Combined With Donafenib in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-002
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Injections; donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Exploration (Experimental): The first stage is a dose-exploration study of ZG005 combined with Donafenib to evaluate the safety and tolerability of different dose combinations in patients with advanced solid tumors who have failed standard therapy.
  Interventions: Drug: ZG005 Powder for Injection; Drug: Donafenib Tosilate Tablets
- Dose Expansion (Experimental): The second stage is a dose-expansion study to further evaluate the safety and initial efficacy of the combination regimen in hepatocellular carcinoma, intrahepatic cholangiocarcinoma, and other potentially beneficial solid tumors.
  Interventions: Drug: ZG005 Powder for Injection; Drug: Donafenib Tosilate Tablets

INTERVENTIONS:
Drug: ZG005 Powder for Injection — intravenous infusion(IV), once every 3 weeks
  Other Names: ZG005
Drug: Donafenib Tosilate Tablets — The dose groups of Donafenib for dose-exploration stage are set as 0.2g BID, 0.1g BID, and 0.1g QD, oral administration.The dose-expansion stage will commence after the Recommended Phase 2 Dose (RP2D) is determined during the dose-escalation stage
  Other Names: Donafenib

SUMMARY:
This is a Multi-center, Open-labe, Phase I/II Study to evaluate the safety and tolerability of ZG005 Combined With Donafenib in Patients With Advanced Solid Tumor.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Male or female 18-70 years of age;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Patients were deemed unsuitable for participating in the study by the investigator for any reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  The sum of the proportions of subjects who achieved CR or PR in imaging evaluation as assessed by the investigator based on RECIST1.1 criteria.
Dose Limiting Toxicity (DLT) | Up to 2 years
  A DLT is defined as any of the following ≥ Grade 3 adverse events occurring from the first dose to the end of first Cycle (21 days), unless the investigator deems that the AE is clearly related to the disease progress or definitely due to an external cause

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 2 years
  Time from the first evaluated CR or PR until PD or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- The Second Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No